CLINICAL TRIAL: NCT01312402
Title: Topical Brinzolamide Ophthalmic Suspension Versus Placebo in the Treatment of Infantile Nystagmus Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Richard W. Hertle, MD, Akron Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101109
Record Dates: First submitted 2011-01-21; First posted 2011-03-10 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Infantile Nystagmus Syndrome
MeSH Terms: interventions — brinzolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical Brinzolamide (Azopt) (Active Comparator): ophthalmic drop given three times a day
  Interventions: Drug: topical brinzolamide 1% in 5mL ophthalmic medication
- placebo ophthalmic drop in 5 mL solution (Placebo Comparator): masked non-active eye drop (absence of Brinzolamide)
  Interventions: Drug: Placebo in 5 mL dispenser

INTERVENTIONS:
Drug: topical brinzolamide 1% in 5mL ophthalmic medication — 1 drop three times a day in both eyes on days 2,3 and 4
  Other Names: Azopt 1% in 5 mL
  Arms: Topical Brinzolamide (Azopt)
Drug: Placebo in 5 mL dispenser — Placebo ophthalmic solution in 5 mL dispenser; 1 drop three times a day on days 2,3 and 4
  Arms: placebo ophthalmic drop in 5 mL solution

SUMMARY:
This study is a prospective, single crossover, double-masked, controlled clinical trial that will use topical brinzolamide (Azopt)ophthalmic medication to try to improve the nystagmus and visual consequences of nystagmus in patients with infantile nystagmus syndrome (INS). Subjects will undergo a clinical exam, questionnaire and eye movement recordings on day 1 and then receive either topical Azopt or placebo three times a day in both eyes for days 2,3 and 4 followed on the morning of day 5 by a repeat clinical exam, questionnaire and eye movement recordings. After at least one week, this protocol is repeated with the crossover regimen being taken by the subject. One week after all medications are discontinued, another clinical exam is done before study discharge. The hypothesis is that nystagmus and associated visual symptoms will be improved while on the Azopt compared to the placebo. There will be a total of 5 visits over a 1-2 month period.

DETAILED DESCRIPTION:
5 subjects are expected to be enrolled in the study. Each subject will be in the study for approximately 1 month.

Efficacy will be assessed by:

* ETDRS Visual Acuity Testing of Binocular Best Corrected Visual Acuity In The Nystagmus Null Zone
* The Validated Amblyopia & Strabismus Ocular Motor Questionnaire
* Eye Movement Recording Data Analysis of The Nystagmus Waveform

Safety will be evaluated by:

* Ocular signs and symptoms
* Visual acuity (uncorrected and best corrected)
* Slit lamp exam and Intraocular Pressure
* Systemic signs and symptoms

ELIGIBILITY:
Inclusion Criteria:

* Age; greater than 12 years old and able to cooperate for full study protocol
* Subject able to understand and sign informed consent
* Subject able to participate in complete ophthalmic and ocular motility evaluation
* Subjects with Infantile Nystagmus Syndrome diagnosed by clinical evaluation and eye movement recordings
* Best-binocular visual acuity in null position 20/50 to 20/200 inclusive using ATS or ETDRS vision testing
* Subject/family able and willing to make the required study visits
* No previous ophthalmic treatment for nystagmus other than for refractive error

Exclusion Criteria:

* Any current use of systemic or topical medications (traditional or non-traditional)
* History of ocular surgery, trauma or chronic ocular disease other than amblyopia
* Systemic diseases requiring medication or other treatments that are known to affect the ocular motor system (e.g., depression, seizure disorders, psychosis)
* Behavioral or neurological disorders which interfere with the study
* Physical or mental impairment precluding study compliance
* Participation in any study involving an IND investigational drug within the past year
* Individual (female) is pregnant, nursing or planning a pregnancy (The safety of Azopt for use during pregnancy has NOT been determined.)
* Periodicity or aperiodicity of INS present on eye movement recordings
* Allergy to sulfa or other components of Azopt solution

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Best Corrected Binocular Visual Acuity | 1 week
  Early Treatment of Diabetic Retinopathy Study Vision Testing Protocol of Best corrected Binocular Acuity

SECONDARY OUTCOMES:
Visual Function | 5 Days
  THe Validated Amblyopia and Visual Function Questionnaire will be administered

CONTACTS AND LOCATIONS:
Overall Officials: Richard W. Hertle, M.D., Principal Investigator — Akron Children's Hospital; Dongsheng Yang, Ph.D., Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

REFERENCES:
- [Background] Dell'Osso LF, Jacobs JB. An expanded nystagmus acuity function: intra- and intersubject prediction of best-corrected visual acuity. Doc Ophthalmol. 2002 May;104(3):249-76. doi: 10.1023/a:1015299930849. PMID 12076015
- [Background] Hertle RW, Dell'Osso LF, FitzGibbon EJ, Thompson D, Yang D, Mellow SD. Horizontal rectus tenotomy in patients with congenital nystagmus: results in 10 adults. Ophthalmology. 2003 Nov;110(11):2097-105. doi: 10.1016/S0161-6420(03)00802-9. PMID 14597515
- [Background] Hertle RW, Anninger W, Yang D, Shatnawi R, Hill VM. Effects of extraocular muscle surgery on 15 patients with oculo-cutaneous albinism (OCA) and infantile nystagmus syndrome (INS). Am J Ophthalmol. 2004 Dec;138(6):978-87. doi: 10.1016/j.ajo.2004.07.029. PMID 15629289
- [Background] Hertle RW, Dell'Osso LF, FitzGibbon EJ, Yang D, Mellow SD. Horizontal rectus muscle tenotomy in children with infantile nystagmus syndrome: a pilot study. J AAPOS. 2004 Dec;8(6):539-48. doi: 10.1016/j.jaapos.2004.08.005. PMID 15616501
- [Background] Jacobs JB, Dell'Osso LF, Hertle RW, Acland GM, Bennett J. Eye movement recordings as an effectiveness indicator of gene therapy in RPE65-deficient canines: implications for the ocular motor system. Invest Ophthalmol Vis Sci. 2006 Jul;47(7):2865-75. doi: 10.1167/iovs.05-1233. PMID 16799026
- [Background] Jacobs JB, Dell'Osso LF, Wang ZI, Acland GM, Bennett J. Using the NAFX to measure the effectiveness over time of gene therapy in canine LCA. Invest Ophthalmol Vis Sci. 2009 Oct;50(10):4685-92. doi: 10.1167/iovs.09-3387. Epub 2009 May 20. PMID 19458334
- [Derived] Hertle RW, Yang D, Adkinson T, Reed M. Topical brinzolamide (Azopt) versus placebo in the treatment of infantile nystagmus syndrome (INS). Br J Ophthalmol. 2015 Apr;99(4):471-6. doi: 10.1136/bjophthalmol-2014-305915. Epub 2014 Oct 21. PMID 25336575